CLINICAL TRIAL: NCT02510807
Title: The PaWS (Pedometer and Walking Study): Comparing Education Alone and Education With Pedometer/Exercise Log Use in Self-monitored Walking in Peripheral Arterial Disease (PAD)
Brief Title: The PaWS (Pedometer and Walking Study)
Acronym: PAWS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: St. Michael (Unknown)
Responsible Party: Principal Investigator, Graham Roche-Nagle, Vascular Surgeon, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-8868-BE
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pedometer group (Experimental): Patients will be instructed to walk a minimum of three times per week up to one half hour total walking time. If they started to get pain in their legs, they will be instructed to stop and rest, and then to start again when the pain has subsided. The pedometer group will be instructed to carry the pedometer in their pocket during these exercise periods.
  Interventions: Other: Pedometer
- Control group (No Intervention): Patients will be instructed to walk a minimum of three times per week up to one half hour total walking time. If they started to get pain in their legs, they will be instructed to stop and rest, and then to start again when the pain has subsided.

INTERVENTIONS:
Other: Pedometer — The use of a pedometer will demonstrate improvement in the following health outcomes in patients with PAD by acting as a method of surveillance to improve compliance with a walking regimen
  Arms: Pedometer group

SUMMARY:
The literature has shown that supervised exercise programs for patients with PAD and who report intermittent claudication (IC) have improved health outcomes, but this is not locally available. Introducing the use of a pedometer may act as a method to encourage patients to continue on their independent exercise regimen. There is very little literature which has examined the effectiveness using pedometers as a measure of compliance within this population.

DETAILED DESCRIPTION:
It has been established that exercise therapy has a central role in the management of peripheral arterial disease. Such treatment should be comprised of intermittent walking of sufficient distance to induce significant discomfort, and be carried out over a period of at least several months. Supervised exercise training utilizing intermittent treadmill walking is a well-validated treatment for claudication. Most prospective randomized single site studies have reported significant improvement in walking distance following supervised exercise training but not with non-supervised regimens.

Furthermore, this has been acknowledged in both the current AHA/ACC 'Guidelines for the management of patients with peripheral arterial disease', which recommends supervised exercise training as an initial treatment modality with a Class 1A level of evidence (highest), as well as in the TransAtlantic Intersocietal Consensus, which provides an 'A' categorical recommendation. In spite of these peer-reviewed, published recommendations, supervised exercise training remains little used, expensive, not reimbursed by Ontario Health Insurance Plan, and therefore is rarely available to patients with claudication in Ontario.

The purpose of this multicentre study is to examine whether the use of a pedometer enhances patient compliance with walking as compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with a diagnosis of PAD (ABI < 0.9) who report symptoms of IC,
* Independent with ambulation (assistive device is permitted) and living independently,
* No previous vascular surgical interventions,
* Fluency in English is preferable but not required,
* Patients need to be willing to return for monthly assessment.

Exclusion Criteria:

* Previous vascular surgical intervention,
* Non-ambulatory,
* Unstable cardiac status (cardiac event < 6 months),
* Cognitive difficulties,
* Unwilling to engage in regular exercise

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Increased walking distance | 6 months
  Six Minute Walk Test
Time to claudication | 6 Months
  Six Minute Walk Test

SECONDARY OUTCOMES:
Quality of Life | 6 months
  ED5QL and the VascuQol-6 questionnaires
Ankle Brachial Index | 6 months
  Ankle Brachial Index
Blood Pressure | 6 months
  Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Graham Roche-Nagle, MD, Principal Investigator — UHN Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fokkenrood HJ, Bendermacher BL, Lauret GJ, Willigendael EM, Prins MH, Teijink JA. Supervised exercise therapy versus non-supervised exercise therapy for intermittent claudication. Cochrane Database Syst Rev. 2013 Aug 23;(8):CD005263. doi: 10.1002/14651858.CD005263.pub3. PMID 23970372
- [Background] Stewart KJ, Hiatt WR, Regensteiner JG, Hirsch AT. Exercise training for claudication. N Engl J Med. 2002 Dec 12;347(24):1941-51. doi: 10.1056/NEJMra021135. No abstract available. PMID 12477945
- [Background] Wind J, Koelemay MJ. Exercise therapy and the additional effect of supervision on exercise therapy in patients with intermittent claudication. Systematic review of randomised controlled trials. Eur J Vasc Endovasc Surg. 2007 Jul;34(1):1-9. doi: 10.1016/j.ejvs.2006.12.030. Epub 2007 Feb 27. PMID 17329131
- [Background] Vemulapalli S, Dolor RJ, Hasselblad V, Schmit K, Banks A, Heidenfelder B, Patel MR, Jones WS. Supervised vs unsupervised exercise for intermittent claudication: A systematic review and meta-analysis. Am Heart J. 2015 Jun;169(6):924-937.e3. doi: 10.1016/j.ahj.2015.03.009. Epub 2015 Mar 26. PMID 26027632
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180